CLINICAL TRIAL: NCT06275880
Title: Effectiveness of Intra-articular Collagen Polyvinylpyrrolidone in Patients With Symptomatic Gonarthross Attended in Rehabilitation of an IMSS-Yucatán Hospital.
Brief Title: Intraarticular Collagen in Patients With Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Roberto Carlos Pech Arguelles, Clinical Professor, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F-2023-3201-066
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Gonarthrosis
Keywords: Gonarthrosis; Collagen; Infiltration
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — collagen-PVP; Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): Patients who received intra-articular infiltration of PVP Collagen
  Interventions: Other: Intra-articular infiltration of PVP Collagen
- GROUP B (Active Comparator): Patients who received conservative treatment through rehabilitation with a home program for one month
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Intra-articular infiltration of PVP Collagen — Intra-articular collagen injection plus physiotherapy program
  Other Names: PVP Collagen
  Arms: GROUP A
Other: Rehabilitation — Patients who received conservative treatment through rehabilitation with a home program for one month
  Arms: GROUP B

SUMMARY:
The objective of this clinical trial is to verify the effectiveness of polyvinyl pyrrolidone collagen in all patients with symptomatic gonarthrosis grades II-IV in patients over 40 years of age. The main objectives that this study aims to answer are the following:

1. - Document the effectiveness of intra-articular polyvinylpyrrolidone collagen in the treatment of symptomatic gonarthrosis.
2. - Compare the intensity of pain, the degree of stiffness and functionality of the joint, prior to application and one month after the therapeutic intervention.
3. - Identify demographic, clinical and therapeutic factors that influence the effectiveness of intra-articular PVP collagen in the treatment of symptomatic gonarthrosis.

Patients diagnosed with symptomatic gonarthrosis Grade II-IV, referred to the Physical Medicine and Rehabilitation service within 3 months, will be selected. Two study groups will be assigned: GROUP those who received intra-articular infiltration of PVP Collagen, GROUP B: patients who received conservative treatment. Through rehabilitation with a home program for one month, in both cases, ENA and the WOMAC scale will be evaluated at the beginning of the study and after 4 weeks.

DETAILED DESCRIPTION:
INTRODUCTION: Osteoarthritis is a disorder characterized by progressive deterioration of cartilage in synovial joints, affecting more than 55% of the elderly population, causing significant physical disability, implying a great challenge in medical treatment.

MATERIAL AND METHODS: A sequential, simple randomized clinical trial was carried out in patients diagnosed with symptomatic gonarthrosis Grade II-IV, referred to the Physical Medicine and Rehabilitation service in 3 months, through two study groups: GROUP Those who received intra-articular infiltration of Collagen PVP, GROUP B: patients who received conservative treatment through rehabilitation with a home program for one month. In both cases, ENA and the WOMAC scale were evaluated at the beginning of the study and at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 40 years.
2. Both sexes.
3. Joint stiffness less than 30 minutes.
4. Crepitus in the knee joint.
5. Pain in one or both knees lasting more than three months.
6. Continuous pain Quantified in >5 Analog Numerical Scale.
7. Patients entitled to the Mexican Social Security Institute.
8. Radiological criteria for gonarthrosis in phases II, III, IV.
9. Patients not candidates for surgical treatment.

Exclusion Criteria:

1. Rheumatoid arthritis, gout or chondrocalcinosis.
2. Treatment with glucosamine, chondroitin, diacerein, silver non-saponifiables or slow-acting drug in the last three months.

4. Anticoagulant treatment. 5. Paget's disease. 6. Treatment with viscosupplementation in the last six months. 7. Patients not entitled to the Mexican Social Security Institute.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index - Pain | One to three months
  number of patients with none, little, quite a bit, a lot, very much
Western Ontario and McMaster Universities Osteoarthritis Index - stiffness | One to Three months
  number of patientes with none, little, quite a bit, a lot, very much
Western Ontario and McMaster Universities Osteoarthritis Index - functionality | One to three months
  number of patients with none, little, quite a bit, a lot, very much
Number Analog Scale for pain | one to three months
  number of patients with 0 (none), 1-2 (very mild pain), 3-4 (mild pain), 5-6 (moderate pain), 7-9 (severe non-disabling pain), 10 (worts pain of life, disabling pain)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Mariela Arriaga Coria, Physician, Principal Investigator — Instituto Mexicano del Seguro Social; Raúl Morales Reyes, Physician, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital General Regional No. 1 Lic. Ignacio García Téllez, Mérida, Yucatán, Mexico

REFERENCES:
- [Background] (1) C. Montoya y Verdugo, Evolución Clínica de los Pacientes con Gonartosis Tratados Mediante la Aplicación de Colágeno de Polivinilpirrolidona, Orthotips Vol. 8 No 2, 2012.
- [Background] (2) M.C. Magaña y Villa, Et Al, Uso de colágeno Polimerizado Tipo I, en el Tratamiento de la Gonartrosis Tipo I, Experiencia en el IMSS, Orthotips. Vol. 8 No 2, 2012.
- [Background] (5) John Richmond, David Hunter et al. Treatment of Osteoarthritis of the Knee, Clinical Practice Guidelines Summary, Journal of the American of Orthopedic Surgeons, 591-600. 2009.
- [Background] (8) Bermúdez Hickey R. Et Al; Tratamiento de la pseudoartrosis de tibia con colágeno polivinilpirrolidona; Rev Mex Ortop Traum 1999; 13(2): 148-151.
- [Background] (9) Campell, C.S. Cirugía Ortopédica. Madrid: Harcourt Brace.
- [Background] (11) Alvarez-López A, Fuentes-Véjar R, Soto-Carrasco SR, Nguyen-Pham T, García-Lorenzo Y de la C, Alvarez-López A, et al. Cartílago y gonartrosis. Revista Archivo Médico de Camagüey [Internet]. 2019 Dec 1;23(6):802-13.
- [Background] (13) Mary O Connor. Sex Difference in Osteoarthritis if the Knee a Hip. Journal of the American of Orthopedic Surgeons, 15; 522-525. 2007.
- [Background] (15) Insall, J.N. Rodilla. New York: Mc. Graw Hill.
- [Background] (16) Salazar-Guzmán I, Garfias- Rosas J, Butze-Rangel W. Mejoria clinica y de la calidad de vida a la aplicación de hialino GF-20 y colageno PVP en pacientes con artrosis de rodilla. Rev Esp Med Quir, 2017;22(1):14-21
- [Background] (20) Laboratorios Aspid S.A. de C.V. Fibroquel® DOF.
- [Background] (22) GPC IMSS-329-10 Evidencias y Recomendaciones. Tratamiento Alternativo en Pacientes con Osteoartrosis de Rodilla Grado I-II
- [Background] (23) M.C. Magaña y Villa, Et Al, Uso de colágeno Polimerizado Tipo I, en el Tratamiento no quirugico de la gonartrosis. Experiencia en el IMSS, Orthotips. Vol. 8 No 2, 2012.
- [Result] Borja-Flores A, Macias-Hernandez SI, Hernandez-Molina G, Perez-Ortiz A, Reyes-Martinez E, Belzazar-Castillo de la Torre J, Avila-Jimenez L, Vazquez-Bello MC, Leon-Mazon MA, Furuzawa-Carballeda J, Torres-Villalobos G, Romero-Hernandez F, Albavera-Hernandez C, Perez-Correa J, Castro-Rocha HA. Long-Term Effectiveness of Polymerized-Type I Collagen Intra-Articular Injections in Patients with Symptomatic Knee Osteoarthritis: Clinical and Radiographic Evaluation in a Cohort Study. Adv Orthop. 2020 Jul 22;2020:9398274. doi: 10.1155/2020/9398274. eCollection 2020. PMID 32802520
- [Result] Jang S, Lee K, Ju JH. Recent Updates of Diagnosis, Pathophysiology, and Treatment on Osteoarthritis of the Knee. Int J Mol Sci. 2021 Mar 5;22(5):2619. doi: 10.3390/ijms22052619. PMID 33807695
- [Result] Watterson JR, Esdaile JM. Viscosupplementation: therapeutic mechanisms and clinical potential in osteoarthritis of the knee. J Am Acad Orthop Surg. 2000 Sep-Oct;8(5):277-84. doi: 10.5435/00124635-200009000-00001. PMID 11029555
- [Result] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Result] Furuzawa-Carballeda J, Rodriquez-Calderon R, Diaz de Leon L, Alcocer-Varela J. Mediators of inflammation are down-regulated while apoptosis is up-regulated in rheumatoid arthritis synovial tissue by polymerized collagen. Clin Exp Immunol. 2002 Oct;130(1):140-9. doi: 10.1046/j.1365-2249.2002.01955.x. PMID 12296865
- [Result] Alvarez-Lopez CA, Garcia-Lorenzo YC. [Relationship between angular deformity and primary osteoarthritis of the knee. Review article]. Acta Ortop Mex. 2015 Jul-Aug;29(4):232-6. Spanish. PMID 27187002
- [Result] Salvatori-Rubi J, Montiel-Jarquin AJ, Lopez-Cazares G, Barragan-Hervella R, Ortiz-Arellano R, Garcia-Carrasco M, Mendoza-Pinto C. [Total knee replacement due to grade IV gonarthrosis]. Acta Ortop Mex. 2014 May-Jun;28(3):193-6. Spanish. PMID 26021117
- [Result] Furuzawa-Carballeda J, Rojas E, Valverde M, Castillo I, Diaz de Leon L, Krotzsch E. Cellular and humoral responses to collagen-polyvinylpyrrolidone administered during short and long periods in humans. Can J Physiol Pharmacol. 2003 Nov;81(11):1029-35. doi: 10.1139/y03-101. PMID 14719037
- [Result] Furuzawa-Carballeda J, Munoz-Chable OA, Macias-Hernandez SI, Agualimpia-Janning A. Effect of polymerized-type I collagen in knee osteoarthritis. II. In vivo study. Eur J Clin Invest. 2009 Jul;39(7):598-606. doi: 10.1111/j.1365-2362.2009.02144.x. Epub 2009 Apr 23. PMID 19397687
- [Result] Furuzawa-Carballeda J, Munoz-Chable OA, Barrios-Payan J, Hernandez-Pando R. Effect of polymerized-type I collagen in knee osteoarthritis. I. In vitro study. Eur J Clin Invest. 2009 Jul;39(7):591-7. doi: 10.1111/j.1365-2362.2009.02154.x. PMID 19453649
- [Result] Furuzawa-Carballeda J, Lima G, Llorente L, Nunez-Alvarez C, Ruiz-Ordaz BH, Echevarria-Zuno S, Hernandez-Cuevas V. Polymerized-type I collagen downregulates inflammation and improves clinical outcomes in patients with symptomatic knee osteoarthritis following arthroscopic lavage: a randomized, double-blind, and placebo-controlled clinical trial. ScientificWorldJournal. 2012;2012:342854. doi: 10.1100/2012/342854. Epub 2012 Apr 1. PMID 22545014
- [Result] Burbano-Levy X, Qf DC, Act EP, Alba IR, Qf LZ. Costo Utilidad de Colagena Polivinil-Pirrolidona en el Tratamiento de Osteartrosis de Rodilla en Mexico. Value Health Reg Issues. 2014 Dec;5:40-47. doi: 10.1016/j.vhri.2014.06.006. Epub 2014 Aug 30. PMID 29702786